CLINICAL TRIAL: NCT05568537
Title: Monitoring Prostate Cancer Tumor Response to Radiation Therapy Using Advanced Functional Magnetic Resonance Imaging (MRI) and Pylarify (18F-DCFPyL) PSMA Positron Emission Tomography (PET)
Brief Title: Prostate MRI and Pylarify PSMA PET/CT
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study withdrawn due to lack of funding and resources
Sponsor: Corewell Health East (Other)
Responsible Party: Principal Investigator, Sirisha Nandalur, MD, Radiation Oncologist, Clinical Faculty, Corewell Health East
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-050
Record Dates: First submitted 2022-09-29; First posted 2022-10-05 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Prostate Cancer
Keywords: MRI; PSMA PET; Pylarify; androgen deprivation therapy; radiation therapy; Pylarify Piflufolastat Flourine-18 (18F-DCFPyL)
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 2-(3-(1-carboxy-5-((6-fluoropyridine-3-carbonyl)amino)pentyl)ureido)pentanedioic acid

STUDY DESIGN:
Intervention Model Description: Non-randomized, prospective, single-institution
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment MRIs and Pylarify PSMA PET/CTs (Experimental): 2 MRIs and 2 Pylarify PSMA PET/CTs, occurring at mid-treatment and when testosterone level is 75% recovered or 12 months after androgen deprivation therapy (ADT), whichever comes first
  Interventions: Drug: Pylarify Piflufolastat Flourine-18 (18F-DCFPyL)

INTERVENTIONS:
Drug: Pylarify Piflufolastat Flourine-18 (18F-DCFPyL) — Piflufolastat F18 will first be given intravenously over about 5 seconds.
  Other Names: Pylarify

SUMMARY:
This is a voluntary research study to find out how using technology including advanced magnetic resonance imaging (MRI) and prostate-specific membrane antigen - positron emission tomography (PSMA-PET) scan imaging, in addition to combined prostate treatment using radiation therapy, brachytherapy (internal radiation treatment using small radioactive seeds placed inside the body) and androgen deprivation therapy (drug therapy to suppress hormones) can help doctors see, track and predict tumor response to treatment for prostate cancer patients. Participation in this study will consist of radiation planning and simulation, magnetic resonance imaging (MRI) and positron emission tomography and computed tomography scan (PET/CT). One MRI and PSMA PET/CT scan will be done prior to the start of first external beam radiation therapy (EBRT) fraction. At mid-treatment prior to the second brachytherapy fraction, an MRI and PSMA PET/CT will be done. A third scan will be performed after 75% testosterone recovery or 12 months post androgen deprivation therapy (ADT) [whichever comes first].

DETAILED DESCRIPTION:
The goal of the study is to better understand how an individual tumor responds to radiation therapy and determine if advanced imaging can be used for prognostic purposes, especially to predict areas of local resistance and failure. The study population are patients with high risk prostate malignancy treated with a combination of external beam radiation therapy (EBRT)/brachytherapy (BT) and androgen deprivation therapy (ADT). Patients enrolled in this trial will undergo a pre-treatment MRI and PSMA PET/CT prior to the initiation of ADT and the first EBRT fraction, a mid-treatment MRI and PSMA PET/CT prior to second brachytherapy fraction, and a third MRI and PSMA PET/CT will be performed after 75% testosterone recovery or 12 months post-ADT (whichever comes first). The pre-treatment MRI and PSMA PET/CT is part of standard of care for prostate cancer workup, however all additional MRI and PSMA PET/CT mid-treatment or after treatment completion are additional research scans.

ELIGIBILITY:
Inclusion Criteria

* Planned definitive radiation for high-risk prostate cancer, radiotherapy plan to include high dose-rate (HDR) brachytherapy boost
* High-risk prostate cancer (tumor stage cT3a-cT4, OR Grade Group 4 or 5, OR prostate-specific antigen (PSA) >20 ng/mL)
* Patients with clinically positive regional lymph nodes
* Patient planned to receive at least 12 months of androgen deprivation therapy
* Age ≥18 years
* No maximum age cutoff, however must have life expectancy > 5 years based on patient's overall health
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Patient able to have 3-Tesla (3T) MRI per Beaumont Radiation Oncology MRI safety questionnaire

Exclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status 3-5
* Metastatic disease
* Prior androgen deprivation therapy before study enrollment
* Prior radiation to pelvis
* Prior malignancy not achieving remission or with prognosis < 5 years
* Synchronous malignancy confirmed or suspected
* Any patient not suitable for brachytherapy
* Severe claustrophobia precluding the acquisition of MRI
* Unable to safely have 3T MRI
* Cognitively impaired

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Difference from baseline (pre-treatment) to mid-treatment scans for each patient in molecular/metabolic MRI to second brachytherapy treatment | From start of treatment to before brachytherapy dose number 2, approximately day 15 of treatment
  Difference in the MRI imaging parameter Amide Proton Transfer (APT) weighted relative signal intensity between pretreatment scan and mid-treatment scan in preselected regions of interest (ROIs) in both high-dose and low-dose regions will be analyzed in each image set per patient.
Difference from baseline (pre-treatment) to end of treatment scans for each patient in molecular/metabolic MRI to second brachytherapy treatment | From start of treatment to 1 year after completion of treatment or recovery of 75% baseline testosterone after androgen depletion therapy.
  Difference in the MRI imaging parameter Amide Proton Transfer (APT) weighted relative signal intensity between pretreatment scan and end-of-treatment scan in preselected regions of interest (ROIs) in both high-dose and low-dose regions will be analyzed in each image set per patient.
Difference from baseline (pre-treatment) to mid-treatment scans for each patient in PSMA PET/CT | From start of treatment to before brachytherapy dose number 2, approximately day 15 of treatment
  Difference in tumor voxel standard uptake value (SUV) between pretreatment scan and mid-treatment scan in preselected regions of interest (ROIs) in both high-dose and low-dose regions will be analyzed in each image set per patient.
Difference from baseline (pre-treatment) to end-of-treatment scans for each patient in PSMA PET/CT | From start of treatment to 1 year after completion of treatment or recovery of 75% baseline testosterone after androgen depletion therapy.
  Difference in tumor voxel standard uptake value (SUV) between pretreatment scan and end-of-treatment scan in preselected regions of interest (ROIs) in both high-dose and low-dose regions will be analyzed in each image set per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Sirisha Nandular, MD, Principal Investigator — Corewell Health East

IPD SHARING:
Plan to Share IPD: No